CLINICAL TRIAL: NCT00800072
Title: Evaluation of NOWOX: a Medical Device Developed to Record Duration of Oxygen Use and Respiration Rate in Patients Requiring Oxygen Therapy
Brief Title: NOWOX Oxygen Therapy Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ALMED-07-MD-015
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: to verify accurrancy of data collected by the NOWOX
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oxygen therapy (Experimental): one experimental device assigned to each of the 10 patients including in the study for an experiemental session duration of 6 hours
  Interventions: Device: NOWOX

INTERVENTIONS:
Device: NOWOX — one experimental device assigned to each of the 10 patients including in the study for an experiemental session duration of 6 hours

SUMMARY:
The purpose of this study is to evaluate the duration of oxygen use recorded by the NOWOX, under usual conditions of daily living, in patients with chronic obstructive respiratory disease requiring oxygen therapy.

DETAILED DESCRIPTION:
Long Term Oxygen Therapy (LTOT) is one of the main non pharmacologic treatments for patients with severe lung disease. This continuous or sub-continuous oxygen supplementation is generally introduced at home in patients who have chronic cardio respiratory failure and severe resting hypoxemia to maintain sufficient blood oxygenation and therefore preserve vital organ function.

LTOT effectiveness has mainly been evaluated and documented in patients with COPD, which also accounts for most of its prescriptions. In these patients, LTOT has been shown to have a beneficial impact on haemodynamics, exercise capacity, lung mechanics and mental state. Its implementation was furthermore associated with reduced yearly hospitalisation days and increased survival Measuring adherence is an extremely important and under-evaluated component of oxygen therapy. NOWOX, medical device has been designed,developed and manufactured to measure adherence to LTOT and additionally to measure patient's respiration rate

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥ 18 years and ≤ 75 years,
* Having a documented diagnosis of moderately severe to severe chronic obstructive respiratory disease
* Hospitalised or out-patient requiring transient or long term oxygen therapy,
* Able to be weaned from oxygen for several consecutive minutes (around 30 minutes, SpO2 at rest on room air should not drop < 85%),
* Able to read
* Willing and able to complete the requirements of this study including providing his/her signature for the written informed consent.

Exclusion Criteria:

* Clinically unstable patient,
* Any contraindication to perform a light cycling exercise, according to the 2003 ATS/ACCP guidelines
* Tracheostomy,
* Nasal obstruction or acute rhinitis occurring in the week prior to selection,
* For female patient:
* Pregnant,
* Positive urinary pregnancy test
* Lactating mother or lack of efficient contraception
* Clinically significant or uncontrolled cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, autoimmune, neurological or psychiatric disorders which may interfere with the study procedures,
* Known allergic reactions to medical material compounds used in the study
* Drug abuse or psychic disorders
* Legal status which prohibits informed consent,
* Participation in any interventional clinical trial within 30 days prior to selection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Primary performance criterion is the overall estimated duration of oxygen use | 6 hours

SECONDARY OUTCOMES:
secondary performance criterion: instantaneous respiration rate recorded by the NOWOX | 6 hours
secondary performance criterion: patient's satisfaction questionnaire on the NOWOX | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Anh-Tuan DINH-XUAN, Professor-MD, Principal Investigator — Department of Physiology - Cochin University Hospital - FRANCE
Locations (1):
- Cochin University Hospital, Paris, France